CLINICAL TRIAL: NCT06786715
Title: Retrograde Intrarenal Surgery (RIRS) With Suction Using Direct in Scope Suction (DISS) Versus Flexible and Navigable Access Sheath (FANS): Randomized Controlled Study
Brief Title: Retrograde Intrarenal Surgery (RIRS) With Suction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Elsayed Abdelhalim Elsayed, assistant lecturer of urology, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFSIRB200-488
Record Dates: First submitted 2025-01-10; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Renal Stone
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Who Masked: Participant
Masking Description: research randomizer
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrograde intrarenal surgery using DISS (Active Comparator): Retrograde intrarenal surgery using DISS
  Interventions: Device: Retrograde intrarenal surgery using DISS
- Retrograde intrarenal surgery using FANS (Active Comparator): Retrograde intrarenal surgery using FANS
  Interventions: Device: Retrograde intrarenal surgery using FANS

INTERVENTIONS:
Device: Retrograde intrarenal surgery using DISS — Retrograde intrarenal surgery using Direct in scope suction for renal stone up to 3 cm
  Arms: Retrograde intrarenal surgery using DISS
Device: Retrograde intrarenal surgery using FANS — Retrograde intrarenal surgery using Flexible and navigable suction for renal stone up to 3 cm
  Arms: Retrograde intrarenal surgery using FANS

SUMMARY:
Suction has been initially used in endoscopic stone management for more than 25 years during PCNL, but the emergence of new devices applying suction through patented ureteroscopes, ureteral access sheaths (UAS) and ureteral catheters led to application of suction in URS/RIRS. The application of ureteral access sheath (UAS) in RIRS can improve surgical vision , reduce intrarenal pressure (IRP) ,and decrease postoperative infectious complications .

ELIGIBILITY:
Inclusion Criteria:

* Single stone
* Medium sized stone ≤ 3 cm
* Renal stone
* age group > 18

Exclusion Criteria:

* multiple renal stones
* stone size > 3 cm
* age group < 18
* solitary kidney
* Obstruction distal to the stone.
* urinary tract infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Stone free rate | One month
  No residual or non siginficant residual less than 4 mm

SECONDARY OUTCOMES:
Operatove data | 2 hours
  Operation and radiation time
Post operative complication | 2 days
  Fever , sepsis , vomitimg

CONTACTS AND LOCATIONS:
Locations (1):
- Elsayed Abdelhalim, Zagazig, Egypt